CLINICAL TRIAL: NCT05057923
Title: The Development of a COVID19 Oral Vaccine Consisting of Bacillus Subtilis Spores Expressing and Displaying the Receptor Binding Domain of Spike Protein of SARS-COV2
Brief Title: The Development of a COVID19 Oral Vaccine Consisting of Bacillus Subtilis Spores
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DreamTec Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRP/008/21FX
Record Dates: First submitted 2021-09-21; First posted 2021-09-27 (Actual); Results first posted 2021-12-23 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Pneumonia
Keywords: Covid-19; Vaccine Reaction; Bacillus subtilis
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: two parallel experimental groups were designed.
  1. the vaccinated volunteers and 2. unvaccinated groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- generation of neutralizing antibody for unvaccinated participants (Experimental): participants received vaccine 1 capsule of 1×10^10 CFU of B. subtilis spore at day 0, 14, and 28 respectively.
  Interventions: Biological: Bacillus subtilis
- neutralizing antibody booster for vaccinated participants (Experimental): participants after 4-month vaccinated with Sinovac received 1 capsule of 1×10^11 CFU of B. subtilis spore
  Interventions: Biological: Bacillus subtilis

INTERVENTIONS:
Biological: Bacillus subtilis — Bacillus subtilis, a harmless intestinal commensal, has earned in recent years, great reputation as a vaccine production host and delivery vector with advantages such as low cost, safe for human consumption and straightforward administration. The technology team has succeeded engineering Bacillus subtilis with spore coat proteins resembling the proteins of the nucleus and spikes of coronal virus. This product could have a vaccine like activity within the intestinal environment.

SUMMARY:
This is a study trial to assess the effectiveness of the immune response stimulated by the genetically engineered Bacillus subtilis which express and display Spike protein of the SARS-COV2 on the spore coat.

DETAILED DESCRIPTION:
Bacillus subtilis is regarded as safe organism by The Food and Drug Administration and it is presented in most food sources. Preliminary experiments have shown that the genetically engineered Bacillus subtilis can express and display receptor binding domain of spike protein of the SARS-COV2 on its spore coat, thus successfully induce the secretion of cytokines of human cells in vitro. Previous experiments also successfully demonstrated that a increased detection of neutralizing IgG and igM levels in mice after oral administrated with the Bacillus subtilis. This suggests that the transgenic spores of Bacillus subtilis have successfully activated the immune system, producing high-affinity neutralizing antibodies and memory B cells. Furthermore, no adverse effects were shown in all the mices. The engineered Bacillus subtilis will be further studied in a human trials through oral administration to test its safety and the immune effect resulted in human bodys.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* age over 25 years
* the outcome of the following examinations should be clinically insignificant: medical and surgical history (hypo-, hypertension, allergy, other diseases, major surgery, micturition, defecation, sleep, illness within the last 4 weeks prior to the start of the trial);
* participant vaccinated with Sinovac over 4 months
* anti-SARS CoV 2 neutralizing antibody is negative in serum.

Exclusion Criteria:

* pregnant women
* history of COVID-19 infection or showing COVID-19 infection symptoms
* having had contact to people with known COVID-19 infection in the last 14 days
* having fever (> 37.4oC in the last 24 hours), dry cough or feeling tired and having aches and pains, nasal congestion, runny nose, sore throat and diarrhea.
* positive real time RT-PCR COVID-19 test.
* persons with autoimmune diseases
* allergic diathesis or any clinically significant allergic disease (i.e. asthma)
* any condition that might impair the immune response
* recent or current immunosuppressive medication
* any other vaccine application 30 days before the first dose

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: WAI YEUNG KWONG, PhD, Principal Investigator — DreamTec Research Limited
Locations (1):
- Zentrogene Bioscience Laboratory Ltd, Hong Kong, Hong Kong

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants voluntary enrolled or recruitted by Genfortune Pharmaceuticals Limited
Pre-assignment Details: 6 unvaccinated participants were recruited and their level of serum neutralizing antibody against spike protein of SARS-CoV2 were lower than 0.003 ug/ml.
Period: Overall Study
Arm/Group | Generation of Neutralizing Antibody for Unvaccinated Participants
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The baseline population does not differ from the participant flow.
Arm/Group | Generation of Neutralizing Antibody for Unvaccinated Participants
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  East Asia | 6

OUTCOME MEASURES:

1. Primary Outcome: Serum Neutralizing Receptor Binding Domain IgG Antibody Concentration
Description: Concentration of neutralizing IgG antibody against receptor binding domain of spike protein in SARS-COV2
Time Frame: Day 0, 27, 42 post oral administration
Population: Participants were orally administered 5x10^7 spores/kg person of recombinant B. subtilis spores mixed with sodium alginate in enteric coated capsules at day 1, 14, and 28. Furthermore, 5 mL of blood samples were drawn at day 0, 27, 42, and the serum samples were analyzed. The titer of neutralizing antibodies was determined with a CLIA-based assay.
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Generation of Neutralizing Antibody for Unvaccinated Participants
Number analyzed (Participants) | 6
ug/ml
  Day 0 | 0.2 (0.1)
  Day 27 | 9.3 (5.4)
  Day 42 | 35.8 (8.8)

2. Secondary Outcome: Lentirival Pseudovirus Neutralization Assay (Wild Type of SARS-CoV2)
Description: The ability of neutralization against SARS-CoV-2 was tested by an in vitro pseudo-virus neutralization assay. The lentivirus carrying a GFP gene was pseudotyped with the spike protein from a wild type of SARS-CoV-2. The pseudoviruses were then pre-incubated with serially diluted serum samples from orally vaccinated volunteers before being added to A549 lung carcinoma cells expressing human ACE2 and human TMPRSS2. The percentage of infection rate was measured with a fluorescent plate reader by counting GFP-positive cells. The results were fitted with a non-linear regression model. The dilution of the serum sample resulted in a 50% reduction of infection rate is designated as EC50. The results were presented as "NA" when the serum samples failed to neutralize pseudovirus infection.
Time Frame: Day 0, 27, 42 post oral administration
Measure: Mean (Standard Deviation); unit: Fold of dilution
Arm/Group | Generation of Neutralizing Antibody for Unvaccinated Participants
Number analyzed (Participants) | 6
Fold of dilution
  EC50 of Day 27 Serum diltuion in Pseudovirus inhibition assay | NA (NA) — The dilution of the serum sample resulted in a 50% reduction of infection rate is designated as EC50. The results were presented as "NA" when the serum samples failed to neutralize pseudovirus infection.
  EC50 of Day 0 Serum diltuion in Pseudovirus inhibition assay | NA (NA) — The dilution of the serum sample resulted in a 50% reduction of infection rate is designated as EC50. The results were presented as "NA" when the serum samples failed to neutralize pseudovirus infection.
  EC50 of Day 42 Serum diltuion in Pseudovirus inhibition assay | 76.33 (38.7)

3. Secondary Outcome: Lentirival Pseudovirus Neutralization Assay (D614G SARS-COV2 Variant)
Description: The ability of neutralization against SARS-CoV-2 was tested by an in vitro pseudo-virus neutralization assay. The lentivirus carrying a GFP gene was pseudotyped with the spike protein from a D614G variant of SARS-CoV-2. The pseudoviruses were then pre-incubated with serially diluted serum samples from orally vaccinated volunteers before being added to A549 lung carcinoma cells expressing human ACE2 and human TMPRSS2. The percentage of infection rate was measured with a fluorescent plate reader by counting GFP-positive cells. The results were fitted with a non-linear regression model. The dilution of the serum sample resulted in a 50% reduction of infection rate is designated as EC50. The results were presented as "NA" when the serum samples failed to neutralize pseudovirus infection.
Time Frame: Day 0, 27, 42 post oral administration
Measure: Mean (Standard Deviation); unit: fold dilution
Arm/Group | Generation of Neutralizing Antibody for Unvaccinated Participants
Number analyzed (Participants) | 6
fold dilution
  EC50 of Day 27 Serum diltuion in Pseudovirus inhibition assay | NA (NA) — The dilution of the serum sample resulted in a 50% reduction of infection rate is designated as EC50. The results were presented as "NA" when the serum samples failed to neutralize pseudovirus infection.
  EC50 of Day 0 Serum diltuion in Pseudovirus inhibition assay | NA (NA) — The dilution of the serum sample resulted in a 50% reduction of infection rate is designated as EC50. The results were presented as "NA" when the serum samples failed to neutralize pseudovirus infection.
  EC50 of Day 42 Serum diltuion in Pseudovirus inhibition assay | 82.4 (29.2)

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected from Day 0 (post-vaccination) up to Day 30 post-final vaccination.
Description: All AEs were presented.
Arm/Group | Generation of Neutralizing Antibody for Unvaccinated Participants
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT05057923/Prot_SAP_ICF_002.pdf